CLINICAL TRIAL: NCT03015779
Title: Transplantation of Autologous Oral Mucosal Epithelial Stem Cell Sheet for Treating Limbal Stem Cell Deficiency Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20161029
Record Dates: First submitted 2017-01-05; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental group (Experimental): cultured autologous oral mucosal epithelial cell sheet
  Interventions: Other: cultured autologous oral mucosal epithelial cell sheet

INTERVENTIONS:
Other: cultured autologous oral mucosal epithelial cell sheet — a prospective study,Before and after self control

SUMMARY:
The aim of this trials investigates the therapeutic effects of application autologous oral mucosal epithelial cell sheets in the treatment of limbal stem cell deficiency disease.

DETAILED DESCRIPTION:
A number of external factors can result in limbal stem cell deficiency(LSCD), causing pain, pathological corneal epithelium regeneration, inflammation reaction and seriously visual loss. For patients with unilaterally damaged eye, transplantation of limbal tissue from the healthy eye can be used in the past years in the risk of inducing limbal stem cell damaged in the healthy eye. While graft of human leukocyte antigen matched allogenic limbal stem cells require immune suppressive medications, it can cause side effects in the body. Over the past 10 years, the clinical trials of application of cultured autologous oral mucosal epithelial cell sheet to treat LSCD have been emerged as a promising strategy in many countries. However, little study has been reported in China. This study investigates the therapeutic effects of application autologous oral mucosal epithelial cell sheets in the treatment of limbal stem cell deficiency disease in China.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged>=18 years old
* Normal intraocular pressure
* Normal Eyelid
* No cataract and retinal disease
* No ulcers and tumor in the mouth

Exclusion Criteria:

* Severe Systemic infection
* History of acute phase of ocular and oral inflammation
* History of hyper sensibility or allergy to antibiotics or serum
* Women who are or may be pregnant
* Patients with infectious diseases
* Patients with other complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The area of reepithelialization of corneal epithelium | 3 months
  The preoperative status of the eye will be recorded on the basis of clinical drawings and pre-and post-operative photographs. These pictures will be sent to two corneal experts in order to evaluate the results.
  Judgement criterion: the results will be tested with a slit lamp:
  Normal: no epithelial loss; Mild: the area of epithelial loss <1/3; Moderate: the area of epithelial loss >1/3 <2/3; Severe: the area of epithelial loss> 2/3

SECONDARY OUTCOMES:
Improvement of best correct visual acuity | one year
Decrease of corneal neovascularization | one year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Zheng Y, Yao T, Wang L, Yu H, Wang Z. Impact of Smoking on the Efficacy of Human Autologous Oral Mucosal Epithelial Cell Sheet Transplantation for Treating Limbal Stem Cell Deficiency. Stem Cells Int. 2026 Jan 5;2026:3769266. doi: 10.1155/sci/3769266. eCollection 2026. PMID 41503585